CLINICAL TRIAL: NCT07357987
Title: Intra-arterial Tenecteplase for Acute Medium Vessel Occlusion Stroke: the ANGEL-MeVO-TNK Randomized Clinical Trial
Brief Title: Intra-arterial Tenecteplase for Acute Medium Vessel Occlusion Stroke
Acronym: ANGEL-MeVO-TNK
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Liping Liu, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANGEL-MeVO-TNK
Record Dates: First submitted 2026-01-11; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Medium Vessel Occlusion; Tenecteplase; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Since the experimental group needs to perform arterial thrombolysis and related operations on patients, the doctors and nurses involved in the study will not be blinded for random patient allocation. However, the grouping of patients will blind neurologists and nurses responsible for conducting neurological, imaging and functional evaluations at baseline and follow-up, as well as collecting clinical outcome data. The randomization information of the patients will also blind the members of the outcome assessment committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IA TNK group (Experimental): During thrombolysis, once vessel recanalization is achieved, immediate termination of the infusion is recommended. If thrombus migration, residual distal embolization, or other situations occur during drug administration, the operator may decide whether to continue treatment at their discretion. Otherwise, TNK will be administered at the specified dose and infusion rate and repeat angiography will be performed after 15 or 30 minutes, followed by termination of the procedure. After completion of the procedure, patients will receive standard medical management as recommended by current guidelines#
  Interventions: Procedure: Intra-arterial Tenecteplase
- Control group (Standard medical management group) (Active Comparator): Patients will receive standard medical management as recommended by current guidelines#
  #《Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke (2023)》and《Chinese Guidelines for Secondary Prevention of Ischemic Stroke and Transient Ischemic Attack (2022)》
  Interventions: Drug: standard medical management

INTERVENTIONS:
Procedure: Intra-arterial Tenecteplase — 1. If the patient has not received IVT, IA TNK will be administered as a slow, continuous infusion at a rate of 0.2-0.3 mg/min for super-selective contact thrombolysis, with a duration of 15-30 minutes. A repeat angiogram will be performed 15 minutes after the start of infusion to assess vessel recanalization, and the operator may decide whether to continue drug administration based on the angiographic findings.
  2. If the patient has received IVT, intra-arterial TNK will be administered as a slow infusion at a rate of 0.2-0.3 mg/min for super-selective contact thrombolysis, with a duration of 15 minutes. For patients with a body weight >80 kg, the infusion rate will be limited to 0.2 mg/min for 15 minutes.
  Arms: IA TNK group
Drug: standard medical management — Patients will receive standard medical management as recommended by current guidelines#
  #《Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke (2023)》and《Chinese Guidelines for Secondary Prevention of Ischemic Stroke and Transient Ischemic Attack (2022)》
  Arms: Control group (Standard medical management group)

SUMMARY:
The ANGEL-MeVO-TNK is a multicentered, prospective, randomized, open label, blinded endpoint (PROBE) phase III trial. A total of 488 AIS patients (age ≥18 years) with acute MeVO-AIS (occlusion of the M2/M3, the A1/A2/A3, the P1/P2/P3, and with baseline NIHSS score >5 or disabling stroke with NIHSS score 3-5 [such as neurological deficits in motor strength, language, vision, etc]), will be enrolled. Patients fulfilling all the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into the IA TNK group or the control group after offering informed content.

* The IA TNK group will receive IA TNK (0.2-0.3 mg/min, for 15 -30min), be infused slowly.
* The control group will be given standard medical management.

The study consists of four visits including the day of randomization, 48±12 hours after randomization, and 90±7 days after randomization. Demographic information, symptoms and signs, laboratory test, neuro-imaging assessment neurological function rating scale will be recorded during the program.

The primary outcome is the modified Rankin Scale (mRS) score of 0 to 1 at 90±7 days after onset. The primary safety outcome is the incidence of sICH within 48±12 hours after randomization (ECASS III).

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria:

1. Age ≥18 years;
2. Pre-stroke mRS 0-1;
3. Within 24 h from symptom onset;
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score >5 or baseline NIHSS 3-5 with disabling deficit (e.g., loss of hand function, aphasia, hemianopia);
5. Informed consent obtained from patients or their legal representatives.

Imaging Inclusion Criteria:

1. Baseline CTA/MRA/DSA diagnosed isolated MeVO, referring to the M2/M3 segment of the MCA, the A1/A2/A3 segment of the ACA, the P1/P2/P3 segment of the PCA;
2. NCCT or MRI DWI imaging showing that the territory of the ischemic infarct volume is less than 50% of the estimated territory supplied by the occluded artery.

Exclusion Criteria:

1. Acute intracranial hemorrhage;
2. ASPECT ≤5;
3. MeVO secondary to spontaneous fragmentation and distal migration of thrombus from an acute large vessel occlusion, or occurring after intravenous thrombolysis (IVT), intra-arterial thrombolysis, or endovascular thrombectomy;
4. Contraindication to TNK;
5. Known severe allergy to contrast agents (excluding mild rash-type allergic reactions);
6. Use of heparin or novel oral anticoagulants within the previous 48 hours with an INR ≥ 1.7;
7. A history of major bleeding within the past 6 months or the presence of conditions such as active gastrointestinal ulcer, aortic dissection, platelet count < 100 × 10⁹/L, etc.;
8. Radiologically confirmed vascular malformations, arterial dissection, intracranial aneurysm (diameter≥3 mm), tumors (except small meningiomas), cerebral vasculitis, cerebral amyloid angiopathy, or other major non-ischemic intracranial diseases (e.g., multiple sclerosis);
9. Acute renal failure, current dialysis, or estimated glomerular filtration rate (eGFR)<30ml/min/1.72m2, and/or serum creatinine>220mmol/L (2.5mg/dl);
10. History of severe liver disease, or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/or glutamyl transferase (GGT) ≥3×upper limit of normal value (ULN) and/or total bilirubin (TBIL) ≥2×ULN;
11. Severe non-cardiovascular comorbidity with an expected life expectancy of less than 3 months (e.g., malignant tumors);
12. Known pregnancy or breastfeeding, or a positive pregnancy test prior to randomization;
13. Current participation in another drug or device clinical trial;
14. Any other condition deemed by the investigator to make the patient unsuitable for participation in the study or to pose a significant risk to the patient (e.g., inability to understand and/or comply with study procedures and/or follow-up due to psychiatric illness, cognitive impairment, or emotional disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
mRS score of 0 to 1 at 90±7 days after onset | 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities, 2 indicating slight disability: unable to carry out all previous activities but able to look after own affairs without assistance; 3 indicating moderate disability: requiring some help, but able to walk without assistance; 4 indicating moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance; 5 indicating severe disability: bedridden, incontinent, and requiring constant nursing care and attention; and 6 indicating death.
symptomatic intracerebral hemorrhage within 48±12 hours after randomization | 48±12 hours after randomization
  symptomatic intracerebral hemorrhage (sICH) within 48±12 hours after randomization (ECASS III criteria)

SECONDARY OUTCOMES:
Ordinal mRS score at 90±7 days after onset | 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities, 2 indicating slight disability: unable to carry out all previous activities but able to look after own affairs without assistance; 3 indicating moderate disability: requiring some help, but able to walk without assistance; 4 indicating moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance; 5 indicating severe disability: bedridden, incontinent, and requiring constant nursing care and attention; and 6 indicating death.
mRS score 0 to 2 at 90±7 days after onset | 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities, 2 indicating slight disability: unable to carry out all previous activities but able to look after own affairs without assistance; 3 indicating moderate disability: requiring some help, but able to walk without assistance; 4 indicating moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance; 5 indicating severe disability: bedridden, incontinent, and requiring constant nursing care and attention; and 6 indicating death.
mRS score 0 to 3 at 90±7 days after onset | 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities, 2 indicating slight disability: unable to carry out all previous activities but able to look after own affairs without assistance; 3 indicating moderate disability: requiring some help, but able to walk without assistance; 4 indicating moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance; 5 indicating severe disability: bedridden, incontinent, and requiring constant nursing care and attention; and 6 indicating death.
Number of Participants with Recanalization of the target occluded artery within 48 ± 12 hours after randomization | 48 ± 12 hours after randomization
  defined as an Arterial Occlusive Lesion [AOL] score of 2-3 on CTA or MRA. The Arterial Occlusive Lesion (AOL) Score is a standardized, angiographic (imaging-based) classification system used to quantify the degree of recanalization (blood flow restoration) in an occluded artery following an endovascular thrombectomy procedure for acute ischemic stroke. Score Range: 0 to 3 (ordinal). A higher score indicates a greater degree of successful mechanical recanalization of the target artery.
Infarct volume at 48 ± 12 hours after randomization | 48 ± 12 hours after randomization
  Infarct volume at 48 ± 12 hours after randomization (assessed by NCCT or MRI DWI)
Change in NIHSS between baseline and 24±2 hours after randomization | 24±2 hours after randomization
  The National Institutes of Health Stroke Scale (NIHSS) is a standardized, quantitative assessment tool used by healthcare providers to objectively evaluate and quantify the neurological deficit and severity of impairment in patients with acute ischemic stroke. Total Score Range: 0 to 42. A higher total score indicates greater neurological impairment.
Number of Participants with Any ICH within 48±12 hours after randomization | 48±12 hours after randomization
  Any ICH within 48±12 hours after randomization
Mortality within 90±7 days after onset | 90±7 days after onset
  Mortality within 90±7 days after onset

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The principal researcher holds complete intellectual property rights. The entire research process and data analysis process strictly protected the information of the subjects. There is not a plan to make individual patient data (IPD) available. Sharing IPD will require IRB approval from Tiantan Hospital and other participating institutes in China.

REFERENCES:
- [Result] Rahme R, Abruzzo TA, Martin RH, Tomsick TA, Ringer AJ, Furlan AJ, Carrozzella JA, Khatri P. Is intra-arterial thrombolysis beneficial for M2 occlusions? Subgroup analysis of the PROACT-II trial. Stroke. 2013 Jan;44(1):240-2. doi: 10.1161/STROKEAHA.112.671495. Epub 2012 Dec 6. PMID 23223507
- [Result] Ospel JM, Menon BK, Demchuk AM, Almekhlafi MA, Kashani N, Mayank A, Fainardi E, Rubiera M, Khaw A, Shankar JJ, Dowlatshahi D, Puig J, Sohn SI, Ahn SH, Poppe A, Calleja A, Hill MD, Goyal M. Clinical Course of Acute Ischemic Stroke Due to Medium Vessel Occlusion With and Without Intravenous Alteplase Treatment. Stroke. 2020 Nov;51(11):3232-3240. doi: 10.1161/STROKEAHA.120.030227. Epub 2020 Oct 19. PMID 33070714
- [Result] Howard G, Waller JL, Voeks JH, Howard VJ, Jauch EC, Lees KR, Nichols FT, Rahlfs VW, Hess DC. A simple, assumption-free, and clinically interpretable approach for analysis of modified Rankin outcomes. Stroke. 2012 Mar;43(3):664-9. doi: 10.1161/STROKEAHA.111.632935. Epub 2012 Feb 16. PMID 22343650
- [Result] Miao Z, Luo G, Song L, Sun D, Chen W, Yao X, Pan Y, Liu Y, Yuan G, Wen C, Wei M, Cai X, Yang Q, Zhou Z, Chang M, Nan G, Wang J, Xiang G, Zhou L, Gao W, Zhang H, Hao J, Xu C, Sun Y, Yi T, Feng G, Han H, Gao F, Ma N, Mo D, Sun X, Deng Y, Tong X, Li X, Jia B, Wang B, He Z, Yang M, Zhao X, Zhang X, Zhang L, Li S, Tong X, Jing J, Xiong Y, Liu T, Li Z, Ren Z, Wang Y, Liebeskind DS, Jovin TG, Nguyen TN, Wang Y, Liu L, Yan B, Huo X; ANGEL-TNK Investigators. Intra-arterial Tenecteplase for Acute Stroke After Successful Endovascular Therapy: The ANGEL-TNK Randomized Clinical Trial. JAMA. 2025 Aug 19;334(7):582-591. doi: 10.1001/jama.2025.10800. PMID 40616323
- [Result] Meng X, Li S, Dai H, Lu G, Wang W, Che F, Geng Y, Sun M, Li X, Li H, Wang Y. Tenecteplase vs Alteplase for Patients With Acute Ischemic Stroke: The ORIGINAL Randomized Clinical Trial. JAMA. 2024 Nov 5;332(17):1437-1445. doi: 10.1001/jama.2024.14721. PMID 39264623
- [Result] Ogawa A, Mori E, Minematsu K, Taki W, Takahashi A, Nemoto S, Miyamoto S, Sasaki M, Inoue T; MELT Japan Study Group. Randomized trial of intraarterial infusion of urokinase within 6 hours of middle cerebral artery stroke: the middle cerebral artery embolism local fibrinolytic intervention trial (MELT) Japan. Stroke. 2007 Oct;38(10):2633-9. doi: 10.1161/STROKEAHA.107.488551. Epub 2007 Aug 16. PMID 17702958
- [Result] Goyal M, Ospel JM, Ganesh A, Dowlatshahi D, Volders D, Mohlenbruch MA, Jumaa MA, Nimjee SM, Booth TC, Buck BH, Kennedy J, Shankar JJ, Dorn F, Zhang L, Hametner C, Nardai S, Zafar A, Diprose W, Vatanpour S, Stebner A, Bosshart S, Singh N, Sebastian I, Uchida K, Ryckborst KJ, Fahed R, Hu SX, Vollherbst DF, Zaidi SF, Lee VH, Lynch J, Rempel JL, Teal R, Trivedi A, Bode FJ, Ogungbemi A, Pham M, Orosz P, Abdalkader M, Taschner C, Tarpley J, Poli S, Singh RJ, De Leacy R, Lopez G, Sahlas D, Chen M, Burns P, Schaafsma JD, Marigold R, Reich A, Amole A, Field TS, Swartz RH, Settecase F, Lenzser G, Ortega-Gutierrez S, Asdaghi N, Lobotesis K, Siddiqui AH, Berrouschot J, Mokin M, Ebersole K, Schneider H, Yoo AJ, Mandzia J, Klostranec J, Jadun C, Patankar T, Sauvageau E, Lenthall R, Peeling L, Huynh T, Budzik R, Lee SK, Makalanda L, Levitt MR, Perry RJ, Hlaing T, Jahromi BS, Singh P, Demchuk AM, Hill MD; ESCAPE-MeVO Investigators. Endovascular Treatment of Stroke Due to Medium-Vessel Occlusion. N Engl J Med. 2025 Apr 10;392(14):1385-1395. doi: 10.1056/NEJMoa2411668. Epub 2025 Feb 5. PMID 39908448
- [Result] Psychogios M, Brehm A, Ribo M, Rizzo F, Strbian D, Raty S, Arenillas JF, Martinez-Galdamez M, Hajdu SD, Michel P, Gralla J, Piechowiak EI, Kaiser DPO, Puetz V, Van den Bergh F, De Raedt S, Bellante F, Dusart A, Hellstern V, Khanafer A, Parrilla G, Morales A, Kirschke JS, Wunderlich S, Fiehler J, Thomalla G, Lemmens R, Peluso JP, Bolognese M, von Hessling A, van Es A, Kruyt ND, Coutinho JM, Castano C, Minnerup J, van Zwam W, Dhondt E, Nolte CH, Machi P, Loehr C, Mattle HP, Buhk JH, Kaesmacher J, Dobrocky T, Papanagiotou P, Alonso A, Holtmannspoetter M, Zini A, Renieri L, Keil F, van den Wijngaard I, Kagi G, Terceno M, Wiesmann M, Amaro S, Rommers N, Balmer L, Fragata I, Katan M, Leker RR, Saver JL, Staals J, Fischer U; DISTAL Investigators. Endovascular Treatment for Stroke Due to Occlusion of Medium or Distal Vessels. N Engl J Med. 2025 Apr 10;392(14):1374-1384. doi: 10.1056/NEJMoa2408954. Epub 2025 Feb 5. PMID 39908430
- [Result] Mohammaden MH, Souza Viana L, Abdelhamid H, Olive-Gadea M, Rodrigo-Gisbert M, Requena M, Martins PN, Matsoukas S, Schuldt BR, Fifi JT, Farooqui M, Vivanco-Suarez J, Ortega-Gutierrez S, Klein P, Abdalkader M, Vigilante N, Siegler JE, Moreira Ferreira F, Peng S, Alaraj A, Haussen DC, Nguyen TN, Nogueira RG. Endovascular Versus Medical Management in Distal Medium Vessel Occlusion Stroke: The DUSK Study. Stroke. 2024 Jun;55(6):1489-1497. doi: 10.1161/STROKEAHA.123.045228. Epub 2024 May 24. PMID 38787927
- [Result] Saber H, Desai SM, Haussen D, Al-Bayati A, Majidi S, Mocco J, Hassan AE, Rajah G, Waqas M, Davies JM, Dornbos D 3rd, Nickele C, Arthur AS, Mowla A, Tenser MS, Mokin M, Pressman E, Aghaebrahim A, Hanel RA, Ortega-Gutierrez S, Jovin T, Duckwiler GR, Liebeskind DS, Nogueira RG, Gornbein J, Saver JL, Jadhav AP. Endovascular Therapy vs Medical Management for Patients With Acute Stroke With Medium Vessel Occlusion in the Anterior Circulation. JAMA Netw Open. 2022 Oct 3;5(10):e2238154. doi: 10.1001/jamanetworkopen.2022.38154. PMID 36279137
- [Result] Guo Y, Wu H, Zhang TY, Li YP, Yang JC, Yang MF, Hu YQ, Zhang HZ. Endovascular treatment achieves better outcomes than best medical management in patients with M2 occlusion and high stroke severity: a meta-analysis. J Neurol. 2023 Jun;270(6):2924-2937. doi: 10.1007/s00415-023-11653-x. Epub 2023 Mar 2. PMID 36862149
- [Result] Duloquin G, Graber M, Garnier L, Crespy V, Comby PO, Baptiste L, Mohr S, Delpont B, Gueniat J, Blanc-Labarre C, Hervieu-Begue M, Osseby GV, Giroud M, Bejot Y. Incidence of Acute Ischemic Stroke With Visible Arterial Occlusion: A Population-Based Study (Dijon Stroke Registry). Stroke. 2020 Jul;51(7):2122-2130. doi: 10.1161/STROKEAHA.120.029949. Epub 2020 Jun 3. PMID 32486967